CLINICAL TRIAL: NCT00456170
Title: Randomized Controlled Trial Comparing Traditional Vaginal Hysterectomy to Harmonic Scalpel Hysterectomy
Brief Title: Are Sutures Required for Vaginal Hysterectomy: A Randomized Controlled Trial
Acronym: HAVE
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Southern Health (Other)
Collaborators: Johnson & Johnson (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Harmonic Vag Hyst
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Vaginal Hysterectomy
Keywords: Vaginal; Hysterectomy; Harmonic; Ligasure; Sutures; Modern; Patients undergoing vaginal hysterectomy for various reasons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Performing Vaginal hysterectomy with Harmonic Scalpel

SUMMARY:
The hypotheses of this study is that the use of the instrument "Harmonic Scalpel" (ultrasonic shears) for vaginal hysterectomy instead of traditional sutures confers advantage over the use of traditional clamps and sutures. The proposed benefits and outcome measures are reduced blood loss, reduced operating time, reduced post-operative pain and earlier discharge from hospital. Other outcome measure will include complications and cost.

DETAILED DESCRIPTION:
Patients booked for vaginal hysterectomy at Southern Health will be offered participation in this trial, and randomised to two separate groups: procedure using ultrasonic shears or traditional sutures. Each patient will receive detailed explanation in document form as well as from the Gynaecology registrar in pre-admission clinic prior to obtaining consent.

After the procedure of vaginal hysterectomy, a research associate will follow these patients up until discharge, collecting relevant data.

A statistician has been employed to perform power calculations, and to analyse data after collection, looking at outcomes mentioned above.

The Harmonic Scalpel has been extensively used to replace the use of traditional clamping and suturing in General Surgery, Laparoscopic surgery, and specifically Total Laparoscopic Vaginal Hysterectomies, but it has never been subjected to a randomised control trial to confirm the anecdotal benefits of the device.

ELIGIBILITY:
Inclusion Criteria:

* Any patient already on waitlist requiring vaginal hysterectomy

Exclusion Criteria:

* No patient consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2007-04

PRIMARY OUTCOMES:
Pain score
Time to discharge
Blood loss

SECONDARY OUTCOMES:
Cost
Complications

CONTACTS AND LOCATIONS:
Overall Officials: Jason J Tan, MBBS MRANZCOG, Principal Investigator — Southern Health
Locations (1):
- Moorabin Hospital, Melbourne, Victoria, Australia